CLINICAL TRIAL: NCT03965884
Title: Investigation of the Effects of Lumbal Stabilization Exercises and Connective Tissue Massage on Neuropathic Pain, Functional Capacity and Quality of Life in Patients With Peripheral Neuropathy
Brief Title: Clinical Effects of Lumbal Stabilization Exercises and Connective Tissue Massage on Neuropathic Pain, Functional Capacity and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, burcu şahin, physiotherapist, Hacettepe University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Neuropathic pain
Record Dates: First submitted 2019-05-12; First posted 2019-05-29 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Physical Therapy Modalities; Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- lumbal stabilization exercise group (Experimental)
  Interventions: Other: Physical therapy and rehabilitation
- connective tissue massage group (Experimental)
  Interventions: Other: Physical therapy and rehabilitation
- control group (No Intervention)

INTERVENTIONS:
Other: Physical therapy and rehabilitation — Physical therapy and rehabilitation
  Arms: connective tissue massage group; lumbal stabilization exercise group

SUMMARY:
The aim of the study is to investigate the efficacy of connective tissue massage and lumbar stabilization exercise treatment on pain severity, functional capacity and quality of life in those who have experienced peripheral neuropathy

DETAILED DESCRIPTION:
The patients diagnosed with fine fiber neuropathy by the neurology department of hacettepe university will be included and the patients referred to physical therapy will be included.

Patients meeting the inclusion criteria will be randomly divided into 3 groups by simple randomization. The first group consisted of lumbal stabilization exercises, the second group with connective tissue massage and the third group with only medical treatment. All patients will be evaluated 2 times before and after 6 weeks. The treatment will be 2 days per week for 6 weeks. Exercise programs of the patients will be performed under the supervision of physiotherapist. In the first group, lumbal stabilization exercises will be applied for 6 weeks and the second group will be given connective tissue massage.

Statistical analysis of the study will be done using SPSS 21 statistical program.

In the statistical analysis to be carried out within the scope of the study, p value will be selected as 0.05 and p <0.05 will be considered significant. Mean ± standard deviation, number, percentage, minimum and maximum values will be used as descriptive statistics. Wilcoxon test is used to compare the pre- and post-treatment values of the groups in the variables and the Kruskal-Wallis test will be used to compare the groups with each other.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed small fiber neuropathy
* Score-4 and over from the -DN4 score
* 18-65 years old adults
* Volunteers to participate in the study.

Exclusion Criteria:

* Pain from different etiologies
* Other neurological disorders involved in neuropathy evaluation
* Cognitive or reading disorders to prevent the questionnaires from being filled
* People with musculoskeletal or orthopedic disorders that affect exercise will not be included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | six week
  visual analogue scale measures pain on a horizontal 100mm line. The most left side on this line is defined no pain and the most right side is defined as 'the most severe pain imaginable'. Patients mark a point on the line according to the pain they feel. The pain level is measured in millimeters from the left to the marked point. we evaluate the current pain, the usual pain in the last month, the worst pain in the last month.

SECONDARY OUTCOMES:
Short Pain Inventory | six week
  Short pain inventory consists of 4 questions evaluating pain severity using number 0 to 10 and 7 questions evaluating the effect of pain on function. The questionnaire requires the patient to consider the current, worst, minimum and mean pain intensity by considering the last week. 0 is defined no pain and 10 is defined as 'the most severe pain imaginable'. Patients are also asked to assess how the pain affects overall activity, walking, normal work, relationships with others, mood, sleep, and enjoyment of life. 0 is defined 'pain has no effect on function', and 10 is defined 'pain has the highest effect on function'.
Neuropathic Pain Impact on Quality of Life questionnaire | six week
  Neuropathic Pain Impact on Quality of Life questionnaire is a self-reported scale used to assess neuropathic pain and its impact on quality of life. The questionnaire contains 42 items in six parameters; psychological, physical, symptoms, personal care, relationships, and social/work activity. The lowest total score that can be obtained from the questionnaire is 42 and the highest score is 210. Increased total score indicates high quality of life
Neuropathic Pain Scale | six week
  Neuropathic Pain Scale is a scale developed to evaluate neuropathic pain quality. The scale includes 2 items that assess the severity of pain and the discomfort of pain, and 8 items that question the character of neuropathic pain. Each item is evaluated with a scale between 0 and 10 points. 0 is defined no pain and 10 is defined as 'the most severe pain imaginable'.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Faculty of Health Sciences Department of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No